CLINICAL TRIAL: NCT02167347
Title: Pilot Study of Culturaly Adapted Family Intervention for Psychosis
Brief Title: Culturally Adapted Family Intervention For Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: University of Manchester (Other); Dow University of Health Sciences (Other); Abbasi Shaheed Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FINT-PSY-02
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Psychosis
Keywords: CBT, Psychosis, cultural adaptation, Pakistan
MeSH Terms: conditions — Psychotic Disorders; Color Vision Defects | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family Intervention (Experimental): Culturally Adapted Family intervention for Psychosis Sessions will be offered weekly basis
  Interventions: Behavioral: Family intervention
- Control (No Intervention): Caregiver ' s Patients who will be randomized to the "treatment as usual" arm will receive routine care

INTERVENTIONS:
Behavioral: Family intervention — This 10 session Multi-modal Psychosocial Intervention will include a supportive component, an educational component, psychosocial component
  Other Names: Psychosocial intervention
  Arms: Family Intervention

SUMMARY:
Aim:

To assess the feasibility of culturally adapted Family Intervention for Psychosis.

Design:

Randomized Control Trial

Setting:

psychiatric department of different hospitals

Participants:

A total of 36 caregivers of Psychosis patients will be randomized to psychological Intervention and treatment as usual arm.

Intervention:

Culturally Adapted Family Intervention for Psychosis

Outcome measure:

Positive and Negative syndrome scale (PANSS) Experience of care -giving inventory(ECI) Care Well-Being & Support(CWS)

DETAILED DESCRIPTION:
The purpose of the study is to test the feasibility of culturally adaptive family intervention for Psychosis

Primary Objective :

* To test whether Pakistani families caring for someone with psychosis will engage with a model of family intervention which has been culturally adapted to meet their needs.
* To evaluate the acceptability of the intervention to the families who receive it and to gather feedback regarding any changes that might improve the intervention.
* To gain an impression of whether the intervention has the potential to address unmet psychological and social needs of the families and how this affects their levels of stress

the investigators will conduct a feasibility pilot study to test whether Pakistani families offered the intervention will want to receive it. The Participants will be recruited from psychiatric department of different hospitals. They will be randomly divided into two groups; intervention group and treatment-as-usual group. A total of thirty six participants will be recruited in the pilot study and divided equally into two arms. This will ensure that, even after loss to follow-up, we will have at least 12 subjects per group for analysis (FDA guidance http://www.fda.gov/cder/guidance/5356fnl.pdf).Randomization will be carried out by the on offsite statistician. This will provide a reliable geographically remote service. For intervention group ten sessions of family intervention will be provided by trained research clinician during the period of three months. Relatives of Patients in the treatment as usual (TAU) group will be given details of intervention at the end of the study and interested families will be offered family intervention

ELIGIBILITY:
Inclusion Criteria:

1. Living with or with at least 10 hours per week face to face contact with an individual with psychosis who has a caring role. Plus the individual with psychosis themselves.
2. Individuals aged between 18-65.
3. Resident of Karachi.
4. Participant is able to give informed written consent.

Exclusion Criteria:

1. Severe drug or alcohol problem (i.e., those who fulfill the criteria for dependence according to ICD10 RDC).
2. Unstable residential arrangements such that the likelihood of being available for the duration of the trial is low.

   .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-02; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Positive and Negative syndrome scale (PANSS) | six months
  The PANSS is a structured clinical interview consisting of 30 items designed to assess severity of symptoms over the past week on a 7-point scale.
Experience of Care-giving inventory(ECI) | six months
  Commonly apply to persons who care for relative or friends With a serious mental illness
Carer Wel-Being & Support(CWS) | six months
  A questionnaire for carers of people with a mental Health problem

SECONDARY OUTCOMES:
Family Questionnaire(FQ) | six months
  Find out the problem of caregiver for relative or friends With a serious mental illness.
Insight rating scale | six months
  Assesses Improvement in insight
Calgary Depression Scale for Schizophrenia | six months
  This is a nine-item scale developed by Addington et al. to assess depression in schizophrenia
Short Explanatory Model Interview | six months
  used to elicit beliefs of mental illness

CONTACTS AND LOCATIONS:
Overall Officials: Nusrat Husain, MD, Principal Investigator — Pakistan Institute of Learning and Living, University of Manchester; Imran Chaudhry, MD, Principal Investigator — University of Manchester; Farooq Naeem, MRCPsych, Principal Investigator — Pakistan Institute of Learning and Living, University of Southampton; Raza Ur Rehman, FCPS, Principal Investigator — Dow University of Health Sciences; Ajmal kazm, Principal Investigator — Pakistan Institute of Living and Learning; Munir Hamirani, FCPS, Principal Investigator — Abbasi Shaheed Hospital
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Husain MO, Khoso AB, Renwick L, Kiran T, Saeed S, Lane S, Naeem F, Chaudhry IB, Husain N. Culturally adapted family intervention for schizophrenia in Pakistan: a feasibility study. Int J Psychiatry Clin Pract. 2021 Sep;25(3):258-267. doi: 10.1080/13651501.2020.1819332. Epub 2020 Sep 15. PMID 32930011